CLINICAL TRIAL: NCT03876899
Title: Evening Primrose Oil for the Treatment of Breastfeeding Related Mastalgia: A Randomized, Double Blinded, Placebo-Controlled Clinical Trial.
Brief Title: RCT of Evening Primrose Oil for the Treatment of Breastfeeding Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLIR 2018-111
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding | interventions — evening primrose oil

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening Primrose Oil (Active Comparator)
  Interventions: Dietary Supplement: Evening Primrose Oil
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Evening Primrose Oil — botanical oil derivative from the seeds of Evening Primrose (Oenothera biennis),1,300 milligrams t.i.d.
  Arms: Evening Primrose Oil
Dietary Supplement: Placebo — Pill
  Arms: Placebo

SUMMARY:
Breastfeeding related mastalgia is a common post-partum complaint. We propose a double-blind, randomized, placebo-controlled trial that investigates the use of Evening Primrose Oil in the treatment of breastfeeding related mastalgia.

ELIGIBILITY:
Inclusion Criteria:

* currently breastfeeding
* recent delivery within the trailing 60 days

Exclusion Criteria:

* history of seizure disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Related Mastalgia | 7 days
  Visual Pain Score

SECONDARY OUTCOMES:
Adverse events | 7 days
  Epistaxis, Change in perceived lochia flow.

IPD SHARING:
Plan to Share IPD: No